CLINICAL TRIAL: NCT00891878
Title: A Randomized Phase II Trial of Sunitinib Plus Capecitabine Versus Capecitabine Alone (With the Potential for Crossover) for Elderly and/or Poor Performance Status Patients With Metastatic Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Capecitabine With or Without Sunitinib Malate as First-Line Therapy in Treating Patients With Metastatic Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0747; NCI-2011-01920 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000641212 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the gastroesophageal junction; recurrent esophageal cancer; stage IV esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Capecitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral capecitabine twice daily on days 1-14. Patients experiencing disease progression may crossover to arm II at the physician's discretion.
  Interventions: Drug: capecitabine
- Arm II (Experimental): Patients receive oral capecitabine as in arm 1 and oral sunitinib malate once daily on days 1-21.
  Interventions: Drug: capecitabine; Drug: sunitinib malate

INTERVENTIONS:
Drug: capecitabine — Given orally
Drug: sunitinib malate — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether capecitabine is more effective when given alone or together with sunitinib malate in treating patients with metastatic esophageal cancer or gastroesophageal junction cancer.

PURPOSE: This randomized phase II trial is studying how well capecitabine works compared with capecitabine given together with sunitinib malate as first-line therapy in treating patients with metastatic cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of elderly (age ≥ 65 years) and/or poor performance status patients with metastatic adenocarcinoma of the esophagus or gastroesophageal junction treated with capecitabine with verus without sunitinib malate.
* Report other indicators of efficacy with these regimens, including the confirmed response rate, overall survival, time to tumor progression, duration of response, and time to treatment failure.
* Compare the adverse event profiles of these regimens in these patients.

Secondary

* Explore whether certain key proteins associated with anti-VEGF therapy are able to predict tumor response.
* Bank paraffin-embedded tissue blocks or slides, and blood products for future studies.

OUTLINE: This is a multicenter study. Patients are stratified according to gender (male vs female), ECOG performance status (0 vs 1 vs 2), and age (≥ 65 years vs < 65 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral capecitabine twice daily on days 1-14. Patients experiencing disease progression may crossover to arm II at the physician's discretion.
* Arm II: Patients receive oral capecitabine as in arm 1 and oral sunitinib malate once daily on days 1-21.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected at baseline for evaluation of protein markers as possible predictors of tumor response to this regimen. Samples are analyzed by IHC for expression levels of markers

After completion of study therapy, patients are followed periodically for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * Metastatic disease
  * Unresectable disease with no curative options
* Measurable disease with ≥ 1 lesion whose longest diameter can be accurately measured as ≥ 2.0 cm by conventional techniques or ≥ 1.0 cm by spiral CT
* Not a candidate for a conventional multi-drug chemotherapy regimen with fairly standard dosing (i.e., patient is able to tolerate at least 80% of standard dosing)

  * Patients who have been offered and declined conventional multi-drug chemotherapy are eligible
* No known CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 and age ≥ 65 years OR PS 2 and age ≥ 18 years but < 65 years
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* Alkaline phosphatase ≤ 2 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60mL/min
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide tissue samples for central review and research purposes
* Able to swallow pills
* No immunocompromised patients (other than related to the use of corticosteroids), including patients known to be HIV-positive
* No co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No NYHA class III or IV heart failure
* No uncontrolled hypertension except at the discretion of treating oncologist
* No other active malignancy except for nonmelanoma skin cancer or carcinoma in situ of the cervix
* No known dihydropyrimidine dehydrogenase deficiency (DPD)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, immunotherapy, or biological therapy for recurrent or metastatic cancer

  * Prior chemotherapy or radiotherapy are allowed if they had been administered as adjuvant or neoadjuvant therapy and a complete surgical resection of the original cancer had been achieved
* No prior sunitinib malate
* No prior radiotherapy to > 30% of the marrow cavity at any time
* More then 4 weeks since prior major surgery
* At least 12 days since prior and no concurrent CYP3A4 inducers, including rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John's wort, efavirenz, and tipranavir
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including azole antifungals (ketoconazole, itraconazole), clarithromycin, erythromycin, diltiazem, verapamil, HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir), and delavirdine
* No other concurrent specific treatment (other than hormonal therapy) in patients with a history of prior malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (182):
- United States (182):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Capecitabine): Patients receive oral capecitabine twice daily on days 1-14. Patients experiencing disease progression may crossover to arm B at the physician's discretion.
- Arm B (Capecitabine+Sunitinib): Patients receive oral capecitabine as in arm 1 and oral sunitinib malate once daily on days 1-21.
Period: Overall Study
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 74.5 [56 to 82] | 73 [47 to 80] | 73 [47 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Progression-free Survival
Description: The primary analysis will be a comparison of Arm A to Arm B using a one-sided log-rank test between the 2 Kaplan-Meier curves. All patients meeting the eligibility criteria, who started treatment will be considered evaluable for the primary endpoint. If a patient is still alive 3 years after registration, no further follow-up is required. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 3 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B (Capecitabine+Sunitinib Malate): Patients receive oral capecitabine as in arm 1 and oral sunitinib malate once daily on days 1-21.
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 6 | 6
Months | 6.1 [0.6 to 9.2] | 2.4 [0.6 to 8.4]
Statistical Analysis 1: Comparison: Arm A (Capecitabine) vs Arm B (Capecitabine+Sunitinib Malate); Test type: Superiority; p = 0.43, Log Rank

2. Secondary Outcome: Response Rate (Complete Response or Partial Response)
Description: A confirmed tumor response is defined to be a CR or PR noted as the objective status on 2 consecutive evaluations ≥4 weeks apart. Confirmed tumor response will be evaluated using the first 6 cycles of treatment. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response. The confirmed response rates between the 2 arms will be compared using a Chi-Square or Fisher's Exact test. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 3 years
Population: All evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 6 | 6
percentage of patients | 0 [0 to 46] | 33 [4 to 78]
Statistical Analysis 1: Comparison: Arm A (Capecitabine) vs Arm B (Capecitabine+Sunitinib Malate); Test type: Superiority; p = 0.45, Fisher Exact

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 6 | 6
Months | 6.2 [1.5 to 18.8] | 5.9 [0.9 to 29.8]

4. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from randomization to the earliest date documentation of disease progression occurs. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of time-to-progression will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 6 | 6
months | 7.56 [1.58 to 9.20] | 2.46 [2.33 to 8.44]

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of randomization to the date at which the patient is removed from treatment due to progression, adverse events, or refusal.
Time Frame: Up to 3 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 6 | 6
months | 1.63 [1.51 to 10.74] | 2.53 [0.69 to 8.48]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Time Frame: Up to 3 years
Population: Patients who achieved an objective response to be either a CR or PR were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Number analyzed (Participants) | 0 | 2
months |  | 4.75 [3.06 to 6.44]

ADVERSE EVENTS:
Arm/Group | Arm A (Capecitabine) | Arm B (Capecitabine+Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Capecitabine) (N=6) | Arm B (Capecitabine+Sunitinib Malate) (N=6)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Capecitabine) (N=6) | Arm B (Capecitabine+Sunitinib Malate) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (29) | 6 (20)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (10) | 2 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (11) | 4 (10)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (3)
Fatigue (General disorders) | 4 (9) | 3 (4)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (9) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (2)
Creatinine increased (Investigations) | 1 (1) | 2 (2)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (9) | 3 (10)
Neutrophil count decreased (Investigations) | 1 (5) | 3 (11)
Platelet count decreased (Investigations) | 1 (1) | 3 (11)
Weight loss (Investigations) | 0 (0) | 1 (8)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (8)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (8) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (8) | 3 (10)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 2 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 2 (3)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (9) | 4 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (4)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes